CLINICAL TRIAL: NCT06384820
Title: A Phase 2 Peri-Operative Study of Treatment With Cemiplimab Alone or in Combination With Fianlimab and/or Other Experimental Agents in Patients With Resectable Stage III/IV Cutaneous Squamous Cell Carcinoma (CSCC)
Brief Title: Study of Cemiplimab Alone or in Combination With Fianlimab and/or Other Experimental Agents in Adult Participants With Peri-operative Stage III/IV Cutaneous Squamous Cell Carcinoma (CSCC)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R3767-ONC-2330; 2023-510514-38-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Cutaneous Squamous Cell Carcinoma
Keywords: Neoadjuvant; Adjuvant; Surgery
MeSH Terms: interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- cemiplimab (Experimental)
  Interventions: Drug: cemiplimab
- fianlimab+cemiplimab (Experimental)
  Interventions: Drug: cemiplimab; Drug: fianlimab

INTERVENTIONS:
Drug: cemiplimab — Administered Intravenous (IV) infusion every three weeks (Q3W)
  Other Names: REGN2810; Libtayo
Drug: fianlimab — IV infusion Q3W
  Other Names: REGN3767
  Arms: fianlimab+cemiplimab

SUMMARY:
This study is researching an investigational drug called REGN2810, also known as cemiplimab, and when combined with another investigational drug called REGN3767, also known as fianlimab (each individually called a "study drug" or called "study drugs" when combined). The study is focused on a type of skin cancer known as cutaneous squamous cell carcinoma (CSCC).

The aim of the study is to see if cemiplimab or cemiplimab in combination with fianlimab can eliminate or reduce the number of living cancer cells in tumor(s) if taken before surgery.

The study is looking at several other research questions, including:

* Whether taking cemiplimab or cemiplimab in combination with fianlimab before surgery may make it possible to have a less extensive surgery or a different treatment plan after surgery
* Whether taking cemiplimab or cemiplimab in combination with fianlimab before surgery may make the cancer less likely to come back after surgery
* What side effects may happen from taking the cemiplimab or cemiplimab in combination with fianlimab
* How much of the cemiplimab or cemiplimab in combination with fianlimab is in the blood at different times
* Whether the body makes antibodies against the study drug(s) (which could make the drug(s) less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Stage III/IV (M0) CSCC, for which surgery would be recommended in routine clinical practice
2. Tumor biopsy is required during screening period as described in the protocol
3. Participant is willing to undergo delayed surgery
4. At least 1 lesion that is measurable by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
6. Adequate organ and bone marrow function as described in the protocol

Key Exclusion Criteria:

1. Stage I or II CSCC
2. Anogenital, penile, vermilion lip CSCC
3. CSCC bone invasion
4. Solid malignancy within 5 years of the projected enrollment date, or hematologic malignancy as described in the protocol
5. Prior radiation therapy for CSCC
6. Myocardial infarction within 6 months of enrollment, or history of myocarditis.
7. Prior treatment with anti-cancer systemic therapy within the last 3 years prior to projected enrollment date as described in the protocol

Note: Other protocol-defined Inclusion/Exclusion Criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11-14 (Estimated); Primary Completion 2026-06-08 (Estimated); Study Completion 2030-05-06 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate by blinded independent pathological review (BIPR) | Up to 100 days

SECONDARY OUTCOMES:
pCR rate by local pathological review | Up to 100 days
Major pathological response (MPR) | Up to 100 days
Event-free survival (EFS) | Up to 3 years
Disease free survival (DFS) | Up to 3 years
Objective response rate (ORR) prior to surgery | Up to 100 days
Overall survival (OS) | Up to 3 years
Occurrence of treatment-emergent adverse events (TEAEs) | Up to 3 years
Occurrence of immune-mediated adverse events (imAEs) | Up to 3 years
Occurrence of treatment-related TEAEs | Up to 3 years
Occurrence of adverse event of special interest (AESI) | Up to 3 years
Occurrence of treatment-emergent serious adverse events (SAEs) | Up to 3 years
Occurrence of laboratory abnormalities | Up to 3 years
  Per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0
Occurrence of death due to TEAE | Up to 3 years
Occurrence of interruption of study drug(s) due to TEAEs | Up to 3 years
Occurrence of discontinuation of study drug(s) due to TEAEs | Up to 3 years
Occurrence of cancellation of surgery due to TEAE | Up to 100 days
Occurrence of delay to surgery due to TEAE | Up to 100 days
Concentrations of cemiplimab in serum | Up to 3 years
Concentrations of fianlimab in serum | Up to 3 years
Concentrations of other experimental agents (as applicable) in serum | Up to 3 years
Incidence of anti-drug antibodies (ADA) to cemiplimab | Up to 3 years
Incidence of ADA to fianlimab | Up to 3 years
Incidence of ADA to other experimental agents (as applicable) | Up to 3 years
Titer of ADA to cemiplimab | Up to 3 years
Titer of ADA to fianlimab | Up to 3 years
Titer of ADA to other experimental agents (as applicable) | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/